CLINICAL TRIAL: NCT05902533
Title: REDEL Trial: Reduced Elective Nodal Dose for Anal Cancer Toxicity Mitigation
Acronym: REDEL
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Jordan Kharofa, Principal Investigator, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCCC-GI-23-01
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Anal Cancer
Keywords: Toxicity Mitigation; Reduced Elective Nodal Dose
MeSH Terms: conditions — Anus Neoplasms | interventions — Radiation; Capecitabine; Mitomycin

STUDY DESIGN:
Intervention Model Description: Single arm prospective trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Reduced Elective Dose + Concurrent Capecitabine/Mitomycin C (Experimental): Reduced elective nodal dose (30.6 Gy); (28- 30 fractions given M-F for approximately 5.5 to 6 weeks) Capecitabine 825 mg/m2 BID on days with RT Mitomycin C 10 mg/m2 slow IV push Days 1 and 29
  Interventions: Radiation: Radiation (reduced elective nodal dose (30.6 Gy); Drug: Capecitabine; Drug: Mitomycin c

INTERVENTIONS:
Radiation: Radiation (reduced elective nodal dose (30.6 Gy) — 28-30 fractions Monday through Friday of intended chemoradiation depending on the total dose required (50.4-54 Gy) which will occur over approximately 5.5 to 6 weeks.
Drug: Capecitabine — 825 mg/m2 BID (Oral Twice daily on days with RT)
Drug: Mitomycin c — 10 mg/m2 slow IV push Day 1 and 29

SUMMARY:
To determine the efficacy of reduced elective nodal radiation in anal cancer patients undergoing chemoradiation in reducing toxicity compared to standard nodal irradiation.

DETAILED DESCRIPTION:
This is a multi-center, single arm prospective trial to evaluate whether reduced elective nodal dose (30.6 Gy) reduces toxicity as defined by the CTCAE Toxicity Index compared to historic patients treated with standard nodal dose on NRG/RTOG0529 and patient reported GI toxicity using the validated PRO-CTCAE scale for diarrhea compared to historic patients treated on UC-GI-1601.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Patients must have stage T1-4N+M0 or T3/T4N0M0 locally advanced anal cancer as evidenced by a PET scan AND either a CT with contrast of the abdomen/pelvis or an MRI with contrast of the pelvis. All imaging must be from within 60 days prior to registration.

   1. Note: Patients with T2N0 disease will be allowed if the primary tumor is >4 cm. Patients with Stage I-T1N0M0 or Stage II-T2N0M0 (tumor ≤ 4cm) will be ineligible for participation.
   2. Patients with perianal cancer that is HPV associated (P16+) will be eligible if the tumor extends to the anal verge and the CTV will include the mesorectal, internal/external iliac, and inguinal lymph nodes.
   3. Patients with excision of the primary tumor but with node positive disease or residual disease at the primary if T3T4N0 will be eligible.
3. ECOG performance status 0 or 1 (or Karnofsky ≥70, see Appendix A).
4. Patients must be able to receive concurrent treatment with capecitabine and Mitomycin C in the opinion of the investigator.
5. Creatinine Clearance must be > 30 ml/min.
6. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Any prior pelvic radiation.
2. History of allergic reactions attributed to compounds of similar chemical or biologic composition to capecitabine.
3. Patients with uncontrolled intercurrent illness that in the opinion of the investigator would prevent receipt of radiation or capecitabine.

   a. Note: HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
4. Pregnant or breastfeeding women are excluded from this study.
5. Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen in the opinion of the investigator.
6. Patients with active autoimmune or connective tissue disease requiring systemic treatment are excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2026-08-14 (Estimated); Study Completion 2029-08-14 (Estimated)

PRIMARY OUTCOMES:
Assess Toxicity Index for all GI, GU, Dermatologic, and Hematologic CTCAE events from treatment initiation through 90 days post treatment | 90 days post treatment
  Toxicity Index for all GI, GU, Dermatologic, and Hematologic CTCAE events from treatment initiation through 90 days post treatment. In patients treated with IMRT enrolled to NRG/RTOG 0529, the mean GI/GU/Derm/Hem TI was 3.858 (SD=0.892) assessed during this time period with standard nodal dose using a simultaneous integrated boost technique. Thirty-three patients will allow an effect size of 0.4 with 80% power and one-sided alpha of 0.05. This effect size is larger than the difference in toxicity observed compared to the historic standard of 3D-conformal radiation with IMRT (current standard) and thus felt to represent a clinically meaningful difference. The CTCAE Toxicity index will be determined for all Dermatologic, Gastrointestinal, Genitourinary, and hematologic events within 90 days from treatment initiation that are possible, probably, or definitely attributable to treatment.
Assess patient reported GI toxicity using PRO-CTCAE Diarrhea | 9 weeks post treatment
  PRO-CTCAE Diarrhea will be used to assess patient reported GI toxicity for the primary endpoint at weeks 3, 5, and 9 (approximately 1-month post-treatment). Any high grade PRO-CTCAE Diarrhea (frequently/almost constantly) in week 3-9 was reported in 71% of patients on a prior trial in this population (UC-GI-1601) with standard nodal dose. With n=33 at alpha =0.05 (actual alpha=0.033) and power=0.80, we can detect a reduction in the proportion of patients reporting any PRO-CTCAE high grade diarrhea (week 3, 5, 9) of at least 22.3%.

SECONDARY OUTCOMES:
Colostomy-Free-Survival - measured by follow up without colostomy | 3 years (Patients followed 3 years post Treatment)
  Colostomy-Free-Survival - Time from treatment completion to any colostomy or last follow up without colostomy.
Disease Free Survival measured by digital rectal exam | 3 and 6 months post treatment
  Disease Free Survival - Failure to achieve complete response (CR) at 6 months or subsequent recurrence. There will be a documented clinical response assessment of the primary anal tumor primarily by using digital rectal exam at 3 and 6 months to define clinical complete response along with a review of imaging at 6 months. Any residual tumor at 6 months would be considered "failure to achieve a complete response" and would be considered a DFS event. Resolution of the primary tumor after chemoradiation and recurrence of tumor (any size) would be considered a DFS event. Persistence of disease in grossly enlarged lymph node (GTV Gross Nodes) at 6 months or resolution and then recurrence (any size) would be considered DFS event. New lesions in the elective nodal space or any other location will be considered a DFS event.
Local Regional Recurrence | 6 months post treatment
  Local Regional Recurrence - All failures within the PTVs for the primary tumor, for the involved Lymph Nodes, or for the Elective Lymph Nodes, including both patients who failed to achieve CR at 6 months and those occurring more than 6 months after completion of chemoradiation after initial CR.
Overall Survival - measured by survival or death at follow up | 3 years (Patients followed 3 years post Treatment)
  Overall Survival - Time from registration to death or last follow up
Proportion of patients requiring a treatment break due to toxicity; measured by more than 3 consecutive fractions missed. | Measured during the 5.5 - 6 week treatment period
  Treatment breaks- The proportion of patients requiring a treatment break due to toxicity (more than 3 consecutive fractions missed) will be monitored and reported. In RTOG 0529, 50% of patients treated with standard nodal dose required a treatment break.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Vermont, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: Undecided